CLINICAL TRIAL: NCT05556018
Title: Activation Pattern and Acute Hemodynamics of His and Left Bundle Pacing
Brief Title: CardioInsight 3 - LBBB
Acronym: CardioInsight3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Bryan Ping Yen YAN, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019.021-T
Record Dates: First submitted 2022-09-16; First posted 2022-09-27 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tailor-made CRT delivery (Experimental): Cardiac resynchronization therapy given according to Electrical Activation Mapping result
  Interventions: Device: Electrical Activation Mapping Guided Cardiac resynchronization therapy

INTERVENTIONS:
Device: Electrical Activation Mapping Guided Cardiac resynchronization therapy — To study the feasibility to optimize configuration of CRT delivery for acute correction of electrical dyssynchrony using a noninvasive mapping of global electrical activation

SUMMARY:
Background Cardiac Resynchronization Therapy (CRT) is proven to improve survival and heart function of patient with certain electrical conduction abnormality and heart failure. However, in patient with certain electrical conduction abnormality, being nonresponder is observed in up to 40% in patient receiving CRT. Conventionally the surgical approach of CRT is to implant one pacing lead in the right heart and one in the left heart to resynchronize the contraction and the pacing lead in the left heart is usually placed in the posterior or lateral portion of the left heart. However, this single approach may not be optimal, especially for those patients with conduction abnormality known to have no response to CRT. Purpose of the clinical investigation The purpose of the Activation Pattern and Acute Hemodynamics of His and Left Bundle Pacing is to study the acute effect on the heart function and conduction abnormality of His and left bundle pacing in conventional CRT candidate. During CRT implantation, Hisbundle lead and Left bundle pacing lead will be placed and the acute effect on heart function will be studied by a wire placed in the left ventricle of the heart and the activation pattern will be studied by a noninvasive global mapping system. The pacing approach that optimally corrects conduction abnormality and improvement on the heart function acutely will be determined

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged 18 or above) of both sexes
* Candidate for CRT therapy according to international guidelines.7
* Informed consent by the patient
* Already received stable dose of guideline directed medical therapy for at least 3 months

Exclusion Criteria:

* Pregnant
* Participating in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2019-07-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in myocardiac activation | 6 months
  Correction of activation abnormality as evaluated by global noninvasive mapping system (ECGi) seen as an increase in acute dp/dt > 5% from baseline with left bundle pacing comparing to biventricular pacing.

SECONDARY OUTCOMES:
Procedure duration | during procedure
  Procedure duration of the optimal CRT delivery method as determined by the best improvement in electrical desynchrony indices.
Implantation success rate | during procedure
  Implantation success rate of the optimal CRT delivery method as determined by the best improvement in electrical desynchrony indices.
Cine images and chest X ray | 6 months
  Cine images (PA, LAO 300, RAO 300) and Chest X ray (PA view) obtained during course of study for assessment of disease
Echocardiogram parameters: strain imaging | 6 months
  Echocardiogram parameters: strain imaging at baseline, 3 months and 6 months
Echocardiogram parameters: left ventricular systolic and diastolic volume | 6 months
  Echocardiogram parameters: left ventricular systolic and diastolic volume at baseline, 3 months and 6 months
Echocardiogram parameters: left ventricular ejection fraction | 6 months
  Echocardiogram parameters: left ventricular ejection fraction at baseline, 3 months and 6 months
Echocardiogram parameters: degree of mitral regurgitation | 6 months
  Echocardiogram parameters at baseline, 3 months and 6 months
Change in New York Heart Association class | 6 months
  Comparison of NYHA class at baseline, 3 months and 6 months to assess changes in quality of life of subject.
Device parameter: defibrillation threshold | 6 months
  Electrical parameters including defibrillation threshold at implant and 6 months follow-up.
post-operative complication rate | 6 months
  Peri-operative and 6 months follow-up complications rate:
  1. Thromboembolic event
  2. Dislodgement and migration of pacing leads
  3. Phrenic nerve stimulation
  4. Others
Device parameter: defibrillation sensitivity | 6 months
  Electrical parameters including defibrillation sensitivity at implant and 6 months follow-up.
Device parameter: lead impedance | 6 months
  Electrical parameters including lead impedance of pacing leads at addition of new lead and 6 months follow-up.
Change in 6 minute hall walk test result | 6 months
  Comparison of 6 minute hall walk test result at baseline, 3 months and 6 months to assess changes in quality of life of subject.
Change in HF Patient Global Assessment Questionnaire outcome | 6 months
  Comparison of HF Patient Global Assessment Questionnaire outcome at baseline, 3 months and 6 months to assess changes in quality of life of subject.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Yan, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong